CLINICAL TRIAL: NCT05648448
Title: ADaptive ASsessment of TReatments for influenzA: A Phase 2 Multi-centre Adaptive Randomised Platform Trial to Assess Antiviral Pharmacodynamics in Early Symptomatic Influenza Infection (AD ASTRA)
Brief Title: A Phase 2 Trial Comparing Antiviral Treatments in Early Symptomatic Influenza
Acronym: AD ASTRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR22003
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-01

CONDITIONS: Influenza; Influenza, Human
Keywords: Influenza; Phase 2; Antiviral Pharmacodynamics
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; favipiravir; Zanamivir; baloxavir; molnupiravir; peramivir; laninamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (11):
- Oseltamivir (TAMIFLU®) (Experimental)
  Interventions: Drug: Oseltamivir
- Favipiravir (Experimental)
  Interventions: Drug: Favipiravir
- Zanamivir (RELENZA®) [Pending addition] (Experimental)
  Interventions: Drug: Zanamivir
- Baloxavir (XOFLUZA®) (Experimental)
  Interventions: Drug: Baloxavir
- Molnupiravir [Pending addition] (Experimental)
  Interventions: Drug: Molnupiravir
- Peramivir (RAPIVAB®) [Pending addition] (Experimental)
  Interventions: Drug: Peramivir
- Laninamivir (INAVIR®) [Pending addition] (Experimental)
  Interventions: Drug: Laninamivir
- Oseltamivir and Baloxavir [Pending addition] (Experimental)
  Interventions: Drug: Oseltamivir and Baloxavir
- Oseltamivir and Favipiravir [Pending addition] (Experimental)
  Interventions: Drug: Oseltamivir and Favipiravir
- Favipiravir and Baloxavir [Pending addition] (Experimental)
  Interventions: Drug: Favipiravir and Baloxavir
- Negative control group (No Intervention): No treatment (except antipyretics- paracetamol)

INTERVENTIONS:
Drug: Oseltamivir — Oral oseltamivir 75mg BD for 5/7
  Arms: Oseltamivir (TAMIFLU®)
Drug: Favipiravir — Oral favipiravir 1800mg BD D0 and 800mg BD for a further 4/7
  Arms: Favipiravir
Drug: Zanamivir — Inhaled zanamivir 10mg BD for 5/7
  Arms: Zanamivir (RELENZA®) [Pending addition]
Drug: Baloxavir — Oral baloxavir:
  * <80kg- single dose of 40mg on D0
  * ≥80kg- single dose of 80mg on D0
  Arms: Baloxavir (XOFLUZA®)
Drug: Molnupiravir — Oral molnupiravir 800mg BD for 5/7
  Arms: Molnupiravir [Pending addition]
Drug: Peramivir — Intravenous peramivir 600mg once only
  Arms: Peramivir (RAPIVAB®) [Pending addition]
Drug: Laninamivir — Inhaled laninamivir 40mg once only
  Arms: Laninamivir (INAVIR®) [Pending addition]
Drug: Oseltamivir and Baloxavir — Oseltamivir 75mg BD for 5/7 and
  Baloxavir:
  * <80kg- single dose of 40mg on D0
  * ≥80kg- single dose of 80mg on D0
  Arms: Oseltamivir and Baloxavir [Pending addition]
Drug: Oseltamivir and Favipiravir — Oseltamivir 75mg BD for 5/7 and
  favipiravir 1800mg BD D0 and 800mg BD for a further 4/7
  Arms: Oseltamivir and Favipiravir [Pending addition]
Drug: Favipiravir and Baloxavir — favipiravir 1800mg BD D0 and 800mg BD for a further 4/7
  Baloxavir:
  * <80kg- single dose of 40mg on D0
  * ≥80kg- single dose of 80mg on D0
  Arms: Favipiravir and Baloxavir [Pending addition]

SUMMARY:
This trial will use a previously validated platform, to quantitatively assess antiviral effects in low-risk patients with high viral burdens and uncomplicated influenza, to determine in-vivo antiviral activity. In this randomised, open-label, controlled, group sequential, adaptive, platform trial, we will compare the performance of available influenza antivirals, and those with potential activity, relative to the control (no treatment) and each other.

AD ASTRA study is supported by the Wellcome Trust Grant ref: 223195/Z/21/Z through the COVID-19 Therapeutics Accelerator

DETAILED DESCRIPTION:
Several influenza antivirals are licensed, differing in availability and routes of administration. Direct comparisons of antiviral and clinical efficacy between the multiple available antivirals are lacking. This comparative information is important for guideline development and for aiding purchasing and prioritisation decisions with several options available.

The platform trial will assess the following interventions:

* Licensed influenza antiviral interventions: oseltamivir (TAMIFLU®), peramivir (RAPIVAB®), zanamivir (RELENZA®), laninamivir (INAVIR®), baloxavir (XOFLUZA®) and favipiravir alone and in combination. The interventions will be chosen in order of priority as well as local feasibility at sites (availability of drugs, local ethics committee and regulatory approvals)
* Interventions with antiviral activity against influenza demonstrated in pre-clinical studies: molnupiravir

Randomisation to the no antiviral treatment control arm (no intervention) will be fixed at a minimum of 20% throughout the study. The randomisation ratios will be uniform for all available interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands the procedures and requirements and is willing and able to give informed consent for full participation in the study
* Adults, male or female, aged 18 to 60 years at time of consent.
* Early symptomatic Influenza (A or B); at least one reported symptom of influenza (including fever, history of fever, myalgias, headache, cough, fatigue, nasal congestion, rhinorrhoea and sore throat) within 4 days (96 hours)
* Influenza positive by rapid antigen test OR a positive RT-PCR test for influenza viruses within the last 24hrs with a Ct value of <30
* Able to walk unaided and unimpeded in activities of daily living (ADLs)
* Agrees and is able to adhere to all study procedures, including availability and contact information for follow-up visits

Exclusion Criteria:

The patient may not enter the study if ANY of the following apply:

* Taking any concomitant medications or drugs which could interact with the study medications or have antiviral activity
* Presence of any chronic illness/condition requiring long term treatment or other significant comorbidity
* BMI ≥35 Kg/m2
* Clinically relevant laboratory abnormalities discovered at screening

  * Haemoglobin <10g/dL
  * Platelet count <100,000/uL
  * ALT > 2x ULN
  * Total bilirubin >1.5 x ULN
  * eGFR <70mls/min/1.73m2
* For females: pregnancy, actively trying to become pregnant or lactation (healthy women on OCP are eligible to join)
* Contraindication to taking, or known hypersensitivity reaction to any of the proposed therapeutics
* Currently participating in another interventional influenza or COVID-19 therapeutic trial
* Clinical evidence of pneumonia- e.g. shortness of breath, hypoxaemia, crepitations (imaging not required)
* Known to be currently co-infected with SARS-CoV-2 (i.e. confirmed with positive ATK or RT-PCR)
* Received live attenuated influenza virus vaccine within 3 weeks prior to study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of viral clearance for currently available drugs and those with potential activity | Days 0 - 5
  Rate of viral clearance- estimated from the log10 viral density derived from qPCR of standardised duplicate oropharyngeal swabs/saliva taken daily from baseline (day 0) to day 7 for each therapeutic arm compared with the no antiviral treatment control i.e. those not receiving study drug

SECONDARY OUTCOMES:
Rate of viral clearance in early influenza infection | Days 0 - 5
  Rate of viral clearance in early influenza infection to characterise the determinants of viral clearance in early influenza infection e.g. contribution of baseline serology, influenza type/subtype, prior vaccination
Rate of viral clearance for drugs shown to have considerable antiviral activity | Days 0 - 5
  Rate of viral clearance for drugs to determine optimal dosing regimens for drugs shown to have considerable antiviral activity
Time to symptom alleviation and fever duration | Days 0 - 14
  Assessment of time to symptom alleviation and fever duration to compare time to symptom resolution and fever duration between interventions

OTHER OUTCOMES:
Rates of hospitalisation for clinical trial reasons | Days 0 - 28
  Rates of hospitalisation for clinical reasons up to day 28
Development of influenza-related complications | Days 0 - 28
  Development of influenza-related complications including bronchitis, sinusitis, otitis media and pneumonia requiring antibiotics, up to day 28
7. Relationship between viral clearance, randomisation arm and other measures (covariates) and development of symptoms or functional issues following illness with influenza. | Days 0-120
  This will be scored using the Modified Influenza Yorkshire Rehabilitation Scale (Flu-YRSm), adapted from the Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm).

CONTACTS AND LOCATIONS:
Locations (4):
- Universidade Federal de Minas Gerais, Minas Gerais, Brazil
- Laos-Oxford-Mahosot Wellcome Trust Research unit, Vientiane, Laos
- Sukraraj Tropical & Infectious Disease Hospital, Kathmandu, Nepal
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With patient's consent, clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future. https://wellcome.ac.uk/press-release/statement-data-sharing-public-health-emergencies).
  The data generated in this study belongs to the study group as a whole. The final database will be shared amongst the site PI and key members of the research team.
  The database may be shared with researchers not directly involved in this study after the main paper has been published and in accordance with MORU guidelines on data sharing.
Access Criteria: Refer to MORU data sharing policy with other researchers to use in the future. https://wellcome.ac.uk/press-release/statement-data-sharing-public-health-emergencies).
URL: http://wellcome.ac.uk/press-release/statement-data-sharing-public-health-emergencies

DOCUMENTS (1):
  • Study Protocol (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT05648448/Prot_002.pdf